CLINICAL TRIAL: NCT05086029
Title: Carpal Tunnel Syndrome in Patients With Psoriatic Arthritis; Superb Microvascular Imaging Findings
Brief Title: Carpal Tunnel Syndrome in Patients With Psoriatic Arthritis
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Ezgi AKYILDIZ TEZCAN, M.D., Selcuk University
Other Study IDs: CTSINPSASMI
Record Dates: First submitted 2021-10-06; First posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Carpal Tunnel Syndrome; Psoriatic Arthritis
Keywords: Carpal Tunnel Syndrome; Psoriatic Arthritis; Superb Microvascular Imaging
MeSH Terms: conditions — Carpal Tunnel Syndrome; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Psoriatic arthritis patients
  Interventions: Diagnostic Test: Superb Microvascular Imaging
- healthy volunteers
  Interventions: Diagnostic Test: Superb Microvascular Imaging

INTERVENTIONS:
Diagnostic Test: Superb Microvascular Imaging — Superb microvascular imaging (SMI) is a new ultrasound technology that can diferen-tiate blood flow signals from artifacts by using a new algorithm.

SUMMARY:
This study aimed to investigate median nerve hypervasculatitation in psoriatic arthritis (PsA) patients with CTS or without CTS by using SMI, then compare them with normal people.

DETAILED DESCRIPTION:
Carpal tunnel syndrome(CTS), a type of median nerve neuropathies, is the most common peripheral nerve entrapment syndrome. Most cases are idiopathic but CTS can be associated with rheumatologic disorders. There isn't any gold standard technique in diagnosis of CTS. Electrodiagnostic studies (EDS) are usually performed to confirm diagnose, to differentiate other diseases or to detect severity. But EDS have some disadvantages such as EDS are time consuming, uncomfortable, may require interventional procedures, can not directly assess the anatomy of the median nerve and its surrounding structures. For these reasons, the use of ultrasonography (US) in the diagnosis of carpal tunnel syndrome has been investigated for a long time. Most of them focused on the cross-sectional area(CSA) of median nerve. Fewer studies have investigated the vascularity of the median nerve. But there is conflict results because conventional Doppler techniques may fail to show small vessels or slow blood flow. Superb microvascular imaging (SMI) is a new ultrasound technology that can diferentiate blood flow signals from artifacts by using a new algorithm. In carpal tunnel syndrome hypervasularitation of median nerve has showed by SMI. To our best knowledge, there isn't any study assessing median nerve hypervascularity by using SMI in PsA. So we aimed to investigate median nerve hypervasculatitation in psoriatic arthritis (PsA) patients with CTS or without CTS by using SMI, then compare them with normal people.

ELIGIBILITY:
Inclusion Criteria:

* PsA patients according to the CASPAR criteria who consecutively applied to the FTR outpatient clinic for PsA follow-up and healthy volunteers who applied to the FTR outpatient clinic enrolled in the study.

Exclusion Criteria:

* Patients were not included in the study if they had a history of wrist or hand fracture, surgery, neurologic disorders such as radiculopathy, polyneuropathy or cerebrovas-cular disease, a history of conditions associated with an increased incidence of CTS such as diabetes mellitus, pregnancy, hypothyroidism or severe systemic diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PsA patients according to the CASPAR criteria who consecutively applied to the FTR outpatient clinic for PsA follow-up and healthy volunteers who applied to the FTR outpatient clinic enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
The blood flow display ratio of SMI in the median nerve | 18 months
  SMI signals will be graded from 0 to 3, in which 0 represented no signal, 1=one to two spot flow, 2= more than two spot flow or one to two strip blood flow (longer than 1 mm) and 3=more than two strip flow

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University Faculty of Medicine, Konya, Turkey (Türkiye)